CLINICAL TRIAL: NCT07357857
Title: Effectiveness of the "High Five!" Program for Reducing the Risk of Overweight and Obesity in Early School-age Children
Brief Title: High Five! - School-based Prevention of Overweight and Obesity Among 6 to 9 Year Olds
Acronym: DINO-PL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mother and Child, Warsaw, Poland (Other)
Collaborators: Ministry of Health, Poland (Other Government)
Responsible Party: Principal Investigator, Prof. Anna Fijałkowska, prof. dr hab. med. i n. o zdr., Institute of Mother and Child, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6/11/85195/NPZ/2021/106/830
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Overweight, Childhood; Obesity Prevention; Blood Pressure
Keywords: children; school-based intervention; overweight prevention; non-communicable diseases prevention; health promotion; health education
MeSH Terms: conditions — Pediatric Obesity; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Students from classes participating in the "High Five!" program (Experimental): High Five!
  Interventions: Behavioral: High Five
- Students from classes not participating in the "High Five!" program (No Intervention): school practice as usual

INTERVENTIONS:
Behavioral: High Five — The "High Five!"program is based on the Life course theory and family-individual-school (FIS) model. Students are the main target groups of the program, and parents cooperate with the school to enhance the effects of the intervention.
  Activities addressed to students include the implementation of 6 scenarios, concerning health-related issues, carried out in accordance with detailed scenarios by trained teacher and school nurse. Parents support th program by performing special home tasks together with the child.
  Arms: Students from classes participating in the "High Five!" program

SUMMARY:
The goal of this interventional study is to assess the effectiveness of the school-based "High Five!" program in reducing overweight, obesity and high blood pressure in children aged 7-9 years old. The main questions it aims to answer are:

* Does participation in the "High Five!" program reduce the proportion of child participants with elevated body mass index (BMI), waist and hip circumference, and blood pressure?
* Does participation in the "High Five!" program increase adherence to recommended health behaviors (healthy eating, physical activity, screen time management, and sleep hygiene) among participating children? Researchers compare "High Five!" to the school practice as usual to see if this program works to prevent overweight and related health problems in children.

Students participate in 6 sessions. Sessions 1-5 are dedicated to five health-related topics such as mental health, nutrition, physical activity, screen time and sleep while session 6 serves as a summarizing and reinforcing lesson. Sessions are based on active methods (play, individual / small group work) and carried out in accordance with detailed scenarios by trained specialists: the class teacher and the school nurse.

Parents/guardians of participating students are engaged in promoting healthy behaviors and creating a supportive home environment via self-reading of the "portions of knowledge" on the topics covered by the program and completion of home tasks with their children.

DETAILED DESCRIPTION:
Background:

Excessive body weight in children is a serious and increasing health problem associated with: elevated blood pressure, risk of obesity in adulthood, poor relationships with peers, negative perception by other (as of lower intelligence, lazy etc.), susceptibility to bullying, low self-esteem and a critical attitude towards oneself.

The key risk factors of overweight in children include: low physical activity, sedentary behaviours, unbalanced diet (too much sugar-sweetened beverages and fast food), sleep disorders and mental health problems.

There are many interventions aimed at reducing overweight and obesity among children, especially those implemented in school settings. However, there is no clear evidence regarding their long-term effectiveness on obesity-related outcomes.

Objectives:

The goal of this clinical trial is to assess the effectiveness of the school-based "High Five!" program in reducing overweight, obesity and high blood pressure in children aged 6-9 years old. The main questions it aims to answer are:

* Does participation in the "High Five!" program reduce the proportion of child participants with elevated body mass index (BMI), waist and hip circumference, and blood pressure?
* Does participation in the "High Five!" program increase adherence to recommended health behaviors (healthy eating, physical activity, screen time management, and sleep hygiene) among participating children?

Intervention:

The High Five! Program is based on the Life course theory claiming that people pass through a sequence of age-based stages and social roles within particular social structures over their lifetime that affects their health, including their body mass. The process of acquiring the skills necessary for living and acting in society to achieve life goals is extremely intensive at the beginning of school, influenced by the social environment. Children learn what behaviors are expected of them and whether they do what they do correctly. Skills acquired at this age and in this environment (classroom) help them cope with new circumstances in the future, thus becoming a lifelong asset. In this context, involving parents in the intervention via assignments, meetings, informative material and encouraging them to improve the home environment is one of the key determinants of the effectiveness of the intervention. In accordance with the family-individual-school (FIS) model of comprehensive childhood obesity prevention, "students connect the family and school, whereas parents collaborate with the school to contribute to the intervention program".

The High Five! Program is adapted to the developmental age of the 7-9 years old participants for whom, play is the favorite form of activity. Children of this age are entering a period of developing perseverance and diligence. Thay want to learn more than ever in their later lives. Therefore, it is extremely important to maintain their enthusiasm and create conditions at school that promote well-being and success. The greatest threat during this period is the child developing a belief in their own low self-worth. Children at this age enjoy listening to and telling stories, which they also use in play. They also enjoy making their own toys. They have good memory skills, especially rhymes and songs. Repetition of the same information promotes memorization. This period is also characterized by the ease of acquiring new motor skills and their improvement. This has a positive impact on daily activities, exercise, participation in sports, crafts, and playing musical instruments. And schoolteachers trained to implement health promoting interventions can have a significant impact on students' dietary behaviors.

The High Five! Program aims to prevent overweight, obesity and high blood pressure in children, by:

* Familiarizing children with health recommendations (eating, sleep, sedentary behaviours, physical activity)
* Strengthening children's skills (positive self-esteem - liking oneself, healthy eating and sleeping, physical activity, screen time control)
* Strengthening the potential of parents to support a healthy lifestyle for their child (modelling of healthy behaviours, encouraging children to follow recommendations, supporting child's positive self-esteem)

The High Five! Program activities include:

* Students participation in 6 sessions. Sessions 1-5 (90 minutes each) are dedicated to five health-related topics:

  1. SUPERPOWERS AND SUPER THOUGHTS- Strengthening positive self-esteem and the ability to see own strengths;
  2. BECOME A CHEF! - Familiarizing children with the current principles of healthy eating and enhance their ability to properly compose meals;
  3. MOVEMENT IS HEALTHY - Familiarize children with the current recommendations for physical activity and motivate them to move ;
  4. TAKE A BREAK - Strengthening motivation and ability to control screen time;
  5. HEALTHY SLEEP - Familiarizing children with the current recommendations for the sleep hours and how to prepare to sleep;
  6. HIGH FIVE FOR HEALTH (45 minutes) - Summarizes and strengthens the program's message in the form of an educational board game.

     Sessions are based on active methods (play, individual / small group work) and carried out in accordance with detailed scenarios by trained specialists: the class teacher and the school nurse.
* Parents' engagement in promoting healthy behaviors and creating a supportive home environment via self-reading of the "portions of knowledge" on the topics covered by the program: mental health, physical activity, nutrition, sleep and screen-time and Completion of home tasks with their children (after the sessions 1-5).

Study design Researchers compare "High Five!" to the school practice as usual to see if this program works to prevent overweight and related health problems in children. The cluster randomized control trial (cRCT) design with a 1:1 ratio (experimental group vs. control group) is applied. The sampling unit is the school, and the sampling is stratified based on the size of the locality (rural/small town/large city). In each school, first- and/or second-grade classes are selected to participate. The characteristics of school environment in terms of systemic/organizational solutions at school that promote healthy eating, physical activity and a social climate friendly to students and parents will be taken into account in the outcome analysis.

Data collection is conducted in four phases: baseline (shortly before the first program session), mid-intervention (in average - after two weeks , post-intervention (shortly after the last program session), and 6-month follow-up. The evaluation includes standardized anthropometric measurements and questionnaires. Children are assessed by school nurses four times, using the Child Examination Report (height, weight, waist/hip circumference, blood pressure). Parents complete a questionnaire evaluating their child's health behaviors (e.g. diet, physical activity, screen time, sleep), emotional well-being (PSC-17), and their own health-related knowledge and supportive parenting practices 3 times (at the baseline, post-intervention and at the follow-up). Students evaluate their own health-related behaviors by marking on the picture scale, for how many days in the last 7 days, they did each of them. They answer the same question four times (at the baseline, mid-intervention, post-intervention, and 6-month follow-up). School staff (e.g., principals) will complete a questionnaire assessing the school's capacity to promote healthy behaviors. This includes food and beverage availability, opportunities for physical activity, school health policies, and implementation of health promotion initiatives.

ELIGIBILITY:
Inclusion Criteria:

Primary schools (public, private, general, inclusive) being a student at a school/class taking part in the study

Exclusion Criteria:

Special schools lack of parental consent for the child to participate in the program lack of child's oral consent to participat

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 659 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the BMI z-score at 6 month | From enrollment to the end of the follow-up at 6 month

SECONDARY OUTCOMES:
Change from Baseline in the percentage of students with values indicating increased Systolic Blood Pressure at 6 Months | From enrollment to the end of the follow-up at 6 month
Change from Baseline in the percentage of students with values indicating increased Diastolic Blood Pressure at 6 Months | From enrollment to the end of the follow-up at 6 month

OTHER OUTCOMES:
Change from baseline in the percentage of students with emotional and behavioral problems based on PSC-17 scores at 6 months | From enrollment to the end of the follow-up at 6 month
  Emotional and behavioral problems in children are assessed by 17-items version of The Pediatric Symptom Checklist (PSC-17) for parents. The total and the subscale scores will be analysed and the following cutoffs will be taken as indicators of the:
  PSC-17 - Inetrnalized problems ≥ 5 PSC-17 - Attention deficites ≥ 7 PSC-17 - Externalized problems ≥7 Total Score ≥ 15
Change from Baseline in the score on the Parental Support and Control scale at 6 Months | From enrollment to the end of the follow-up at 6 month
  The Parental Support and Control 20-items scale was developed specifically for this study. It consists of 20 statements describing parental behaviors that express emotional support for the child (10 statements, e.g. "I hug and cuddle my child") and control of the child (10 statements, e.g. "I know my child's friends"). For each statement, respondents select one of the following answers: 0 - "Rarely"; 1 - "Sometimes"; 2 - "Often". The higher the score, the stronger the support and control of the child by the parents.
  Both the subscale scores and the overall score will be analyzed. Since the scale was previously only pilot tested in a small group, the analysis of its psychometric properties will precede the analysis of the program results.
Change from baseline in the percentage of students meeting recommendations for daily moderate physical activity (MVPA) after 6 months | From enrollment to the end of the follow-up at 6 months
  The assessment is based on parents' answer to the single question on the numer of days per week the child meets the WHO recommendation for daily MVPA (Moderate-to-Vigorous Physical Activity) - being active for at least 60 minutes.
Change from baseline in the percentage of students regularly (at least 3-4 hours per week) attending sports clubs | From enrollment to the end of the follow-up at 6 months
  Assessment based on parental responses to the question, "In a typical week (including weekends), how much time does your child spend on average playing sports/exercise/dance classes at a sports club/health club/fitness center/dance academy? (By sports and exercise, we mean soccer, playing on the field, hockey, swimming, tennis, basketball, gymnastics, ballet, fitness classes, dance classes, etc.)." 5-point response scale: Not at all; 1-2 hours per week; 3-4 hours per week; At least 5 hours per week; I don't know
Change from baseline in the percentage of students who regularly and actively participate in sports | From enrollment to the end of the follow-up at 6 months
  Assessment based on parental responses to the question "Does your child participate in sports club activities?" 4-point response scale: Yes, regularly and actively; Yes, occasionally; Not currently, but has participated in the past; No and has never participated
Change in the percentage of students sleeping for at least 9 hours per day compared to baseline. | From enrollment to the end of the follow-up at 6 months
  The child's sleep time is assessed by parents who indicate the time a child usually falls asleep (hours and minutes) and the time child usually wakes-up (hours and minutes).
Change from baseline in the percentage of students who regularly (every day) eat breakfast | From enrollment to the end of the follow-up at 6 months
  Parents answer the question: "In a typical week, how often does your child eat breakfast (something more than just a drink, e.g., milk, tea, juice), including breakfast at school? Please select one answer. Never; A few days (1-3 days); Most days (4-6 days); Every day
Change from baseline in the percentage of students meeting WHO recommendations for daily fruit and vegetable consumption (at least 5 servings per day) | From enrollment to the end of the follow-up at 6 months
  Parents answer the question: "In a typical week, how many servings of fresh fruit and/or vegetables does your child eat per day? (One serving is the amount your child can fit in the palm of their hand, e.g., 4 dessert spoons of cooked vegetables, a small bowl of salad, a small bowl of vegetable soup; 1 medium-sized fruit [1 small apple], 2 small fruits [2 plums], 4-7 strawberries, or 10-14 cherries.)" choosing one of the categories: Not at all; Less than 1 serving per day; 1-2 servings per day; 3-4 servings per day; 5 or more servings per day
Change from baseline in the mean number of hygiene rules related to nighttime rest and the preparation to it regularly (5-7 day per week) followed by children | From enrollment to the end of the follow-up at 6 months
  The index of rules for good sleep for children is composed of five questions answered by parents and covers: bathing/showering, brushing teeth, airing the room, relaxation (listening to a bedtime story, talking with a parent, etc.) before bad and not watching TV or using a cell phone for at least half an hour before bed. For each question, parents can choose one of three answers: (Usually (5-7 days a week); Sometimes (2-4 days a week); Rarely (1-2 days a week)) and the indicator of regular use of a given practice is the answer "Usually (5-7 days a week)"
Change from baseline in the percentage of students who regularly consume fresh fruits. | From enrollment to the end of the follow-up at 6 months
  Parents indicated how often, considering a typical week, their child consumes fresh fruit (excluding fruit juices and dried fruit) choosing one out of six response categories ranging from Never to More than once a day. Responses ranging from Once a day to More than once a day indicate regular consumption.
Change from baseline in the percentage of students who regularly consume vegetables. | From enrollment to the end of the follow-up at 6 months
  Parents indicated how often, considering a typical week, their child consumes vegetables (including vegetable soups, excluding potatoes) choosing one out of six response categories ranging from Never to More than once a day. Responses ranging from Once a day to More than once a day indicate regular consumption.
Change from baseline in the percentage of students who frequently consume sugar-containing beverages | From enrollment to the end of the follow-up at 6 months
  Parents indicated how often, considering a typical week, their child consumes sugar-containing beverages choosing one out of six response categories ranging from Never to More than once a day. Responses ranging from 4 to 6 - more than 3 days per week indicate frequent consumption.
Change from baseline in the percentage of students who frequently consume salty snacks | From enrollment to the end of the follow-up at 6 months
  Parents indicated how often, considering a typical week, their child consumes salty snacks (e.g. potato chips, corn chips, popcorn, peanuts) choosing one out of six response categories ranging from Never to More than once a day. Responses ranging from 4 to 6 - more than 3 days per week indicate frequent consumption.
Change from baseline in the percentage of students who frequently consume sweet snacks | From enrollment to the end of the follow-up at 6 months
  Parents indicated how often, considering a typical week, their child consumes sweet snacks (e.g. cakes, cookies/biscuits, sweet desserts) choosing one out of six response categories ranging from Never to More than once a day. Responses ranging from 4 to 6 - more than 3 days per week indicate frequent consumption.
Change from baseline in the percentage of students who frequently consume fast food products | From enrollment to the end of the follow-up at 6 months
  Parents indicated how often, considering a typical week, their child consumes fast food products (e.g. pizza, casserole, hamburger) choosing one out of six response categories ranging from Never to More than once a day. Responses ranging from 4 to 6 - more than 3 days per week indicate frequent consumption.
Change from baseline in the percentage of students who regularly (daily) eat breakfast with at least one parent. | From enrollment to the end of the follow-up at 6 months
  Parents indicate how often, on a typical week, they eat breakfast with a child by choosing one of the answers: Never, Less than once a week, 1-2 days a week, 3-4 days a week, 5-6 days a week, Every day. Two last categories indicate regular behavior.
Change from baseline in the percentage of students who regularly (daily) eat lunch with at least one parent | From enrollment to the end of the follow-up at 6 months
  Parents indicate how often, on a typical week, they eat lunch with a child by choosing one of the answers: Never, Less than once a week, 1-2 days a week, 3-4 days a week, 5-6 days a week, Every day. Two last categories indicate regular behavior.
Change from baseline in the percentage of students who regularly (daily) eat diner with at least one parent | From enrollment to the end of the follow-up at 6 months
  Parents indicate how often, on a typical week, they eat diner with a child by choosing one of the answers: Never, Less than once a week, 1-2 days a week, 3-4 days a week, 5-6 days a week, Every day. Two last categories indicate regular behavior.
Change from baseline in the average time spent by students on playing games on a computer, console, tablet, smartphone, TV | From enrollment to the end of the follow-up at 6 months
  Parents answer the question "In their free time: how many hours a day does your child spend on playing games on a computer, console, tablet, smartphone, TV" by selecting one of 9 answers (from Not at all to About 7 or more hours a day)
Change from baseline in the average time spent by students using a computer or other electronic devices for academic activities, including homework | From enrollment to the end of the follow-up at 6 months
  Parents answer the question "In their free time: how many hours a day does your child spend using a computer or other electronic devices for academic activities, including homework" by selecting one of 9 answers (from Not at all to About 7 or more hours a day)
Change from baseline in the average time spent by students on watching TV, movies or videos on sites like YouTube, etc. | From enrollment to the end of the follow-up at 6 months
  Parents answer the question "In their free time: how many hours a day does your child spend watching TV, movies or videos on sites like YouTube, etc." by selecting one of 9 answers (from Not at all to About 7 or more hours a day)
Change from baseline in the average time spent by students searching for information on the Internet, browsing websites | From enrollment to the end of the follow-up at 6 months
  Parents answer the question "In their free time: how many hours a day does your child spend searching for information on the Internet, browsing websites." by selecting one of 9 answers (from Not at all to About 7 or more hours a day)
Change from baseline in the average time spent by students on other sedentary activities, e.g. reading books, playing an instrument | From enrollment to the end of the follow-up at 6 months
  Parents answer the question "In their free time: how many hours a day does your child spend on other sedentary activities, e.g. reading books, playing an instrument." by selecting one of 9 answers (from Not at all to About 7 or more hours a day)
Change from baseline in the average number of days in the past seven days students consumed vegetables | From enrollment to the end of the follow-up at 6 months
  Students mark on the picture scale answer to the question "How many days in the last week (last 7 days) did you eat vegetables - fresh (e.g., carrots) or cooked (e.g., broccoli, potatoes)?". They select one out of five answers: never, 1 day, 2-3 days, 4-5 days, 6-7 days
Change from baseline in the average number of days in the past seven days students consumed fruits | From enrollment to the end of the follow-up at 6 months
  Students mark on the picture scale answer to the question: "How many days in the last week (last 7 days) did you eat fruit - for example, an apple, a banana or a pear?". They select one out of five answers: never, 1 day, 2-3 days, 4-5 days, 6-7 days
Change from baseline in the average number of days in the past seven days students actively commuted to/from school | From enrollment to the end of the follow-up at 6 months
  Students mark on the picture scale answer to the question: "How many days in the last week (last 7 days) did I walk, ride a bike, ride a scooter to (or from) school?". They select one out of five answers: never, 1 day, 2-3 days, 4-5 days, 6-7 days
Change from baseline in the average number of days in the past seven days students were physically active | From enrollment to the end of the follow-up at 6 months
  Students mark on the picture scale answer to the question: "How many days in the last week (last 7 days) you were active - you moved a lot, ran, danced, played football or swam?" They select one out of five answers: never, 1 day, 2-3 days, 4-5 days, 6-7 days
Change from baseline in the average number of days in the past seven days students slept for 9 hours or more | From enrollment to the end of the follow-up at 6 months
  Students mark on the picture scale answer to the question: "How many days in the last week (last 7 days) you slept for 9 hours or more last night?" They select one out of five answers: never, 1 day, 2-3 days, 4-5 days, 6-7 days
Change from baseline in the average number of days in the past seven days students calmed down before going to bed | From enrollment to the end of the follow-up at 6 months
  Students mark on the picture scale answer to the question: "How many days in the last week (last 7 days) before going to bed, you listened to calming music, a story, or read something interesting?" They select one out of five answers: never, 1 day, 2-3 days, 4-5 days, 6-7 days
Change from baseline in the average number of days in the past seven days students spent less than 2 hours in front of the computer, phone, or tablet. | From enrollment to the end of the follow-up at 6 months
  Students mark on the picture scale answer to the question: "How many days in the last week (last 7 days) did you spent less than 2 hours in front of the computer, phone, or tablet?" They select one out of five answers: never, 1 day, 2-3 days, 4-5 days, 6-7 days
Change from baseline in the average number of days in the past seven days students did not use the phone, computer, or tablet right before going to bed | From enrollment to the end of the follow-up at 6 months
  Students mark on the picture scale answer to the question: "How many days in the last week (last 7 days) you did not use the phone, computer, or tablet right before going to bed?" They select one out of five answers: never, 1 day, 2-3 days, 4-5 days, 6-7 days
Change from baseline in the average number of days in the past seven days students played with other children outdoor after school | From enrollment to the end of the follow-up at 6 months
  Students mark on the picture scale answer to the question: "How many days in the last week (last 7 days) after school you played with other children, e.g., in the yard or on the playground?" They select one out of five answers: never, 1 day, 2-3 days, 4-5 days, 6-7 days
Change from baseline in the average number of days in the past seven days students spent free time with their loved ones | From enrollment to the end of the follow-up at 6 months
  Students mark on the picture scale answer to the question: "How many days in the last week (last 7 days) did you spent free time with your loved ones - you played together, talked, or did something else?" They select one out of five answers: never, 1 day, 2-3 days, 4-5 days, 6-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Anna Fijałkowska, Professor, Principal Investigator — Institute of Mother and Child
Locations (1):
- Institute of Mother and Child, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao ZJ, Wang SM, Chen Y. A randomized trial of multiple interventions for childhood obesity in China. Am J Prev Med. 2015 May;48(5):552-60. doi: 10.1016/j.amepre.2014.12.014. PMID 25891054
- [Background] Wang Y, Cai L, Wu Y, Wilson RF, Weston C, Fawole O, Bleich SN, Cheskin LJ, Showell NN, Lau BD, Chiu DT, Zhang A, Segal J. What childhood obesity prevention programmes work? A systematic review and meta-analysis. Obes Rev. 2015 Jul;16(7):547-65. doi: 10.1111/obr.12277. Epub 2015 Apr 20. PMID 25893796
- [Background] Telama R. Tracking of physical activity from childhood to adulthood: a review. Obes Facts. 2009;2(3):187-95. doi: 10.1159/000222244. Epub 2009 Jun 12. PMID 20054224
- [Background] Smit MS, Boelens M, Molenberg FJM, Raat H, Jansen W. The long-term effects of primary school-based obesity prevention interventions in children: A systematic review and meta-analysis. Pediatr Obes. 2023 Mar;18(3):e12997. doi: 10.1111/ijpo.12997. Epub 2022 Dec 21. PMID 36545748
- [Background] Sluggett L, Wagner SL, Harris RL. Sleep Duration and Obesity in Children and Adolescents. Can J Diabetes. 2019 Mar;43(2):146-152. doi: 10.1016/j.jcjd.2018.06.006. Epub 2018 Jul 4. PMID 30266216
- [Background] Simmonds M, Llewellyn A, Owen CG, Woolacott N. Predicting adult obesity from childhood obesity: a systematic review and meta-analysis. Obes Rev. 2016 Feb;17(2):95-107. doi: 10.1111/obr.12334. Epub 2015 Dec 23. PMID 26696565
- [Background] Rousham EK, Goudet S, Markey O, Griffiths P, Boxer B, Carroll C, Petherick ES, Pradeilles R. Unhealthy Food and Beverage Consumption in Children and Risk of Overweight and Obesity: A Systematic Review and Meta-Analysis. Adv Nutr. 2022 Oct 2;13(5):1669-1696. doi: 10.1093/advances/nmac032. PMID 35362512
- [Background] Lambrinou CP, Androutsos O, Karaglani E, Cardon G, Huys N, Wikstrom K, Kivela J, Ko W, Karuranga E, Tsochev K, Iotova V, Dimova R, De Miguel-Etayo P, M Gonzalez-Gil E, Tamas H, Jancso Z, Liatis S, Makrilakis K, Manios Y; Feel4Diabetes-study group. Effective strategies for childhood obesity prevention via school based, family involved interventions: a critical review for the development of the Feel4Diabetes-study school based component. BMC Endocr Disord. 2020 May 6;20(Suppl 2):52. doi: 10.1186/s12902-020-0526-5. PMID 32370795
- [Background] Kulaga Z, Swiader-Lesniak A, Kotowska A, Litwin M. Population-based references for waist and hip circumferences, waist-to-hip and waist-to-height ratios for children and adolescents, and evaluation of their predictive ability. Eur J Pediatr. 2023 Jul;182(7):3217-3229. doi: 10.1007/s00431-023-05001-4. Epub 2023 May 4. PMID 37140701
- [Background] Jebeile H, Kelly AS, O'Malley G, Baur LA. Obesity in children and adolescents: epidemiology, causes, assessment, and management. Lancet Diabetes Endocrinol. 2022 May;10(5):351-365. doi: 10.1016/S2213-8587(22)00047-X. Epub 2022 Mar 3. PMID 35248172
- [Background] Jakobsen DD, Brader L, Bruun JM. Association between Food, Beverages and Overweight/Obesity in Children and Adolescents-A Systematic Review and Meta-Analysis of Observational Studies. Nutrients. 2023 Feb 2;15(3):764. doi: 10.3390/nu15030764. PMID 36771470
- [Background] Habib-Mourad C, Ghandour LA, Maliha C, Awada N, Dagher M, Hwalla N. Impact of a one-year school-based teacher-implemented nutrition and physical activity intervention: main findings and future recommendations. BMC Public Health. 2020 Feb 19;20(1):256. doi: 10.1186/s12889-020-8351-3. PMID 32075607
- [Background] Cockerham WC. Theoretical Approaches to Research on the Social Determinants of Obesity. Am J Prev Med. 2022 Jul;63(1 Suppl 1):S8-S17. doi: 10.1016/j.amepre.2022.01.030. PMID 35725145
- [Background] Calcaterra V, Cena H, Magenes VC, Vincenti A, Comola G, Beretta A, Di Napoli I, Zuccotti G. Sugar-Sweetened Beverages and Metabolic Risk in Children and Adolescents with Obesity: A Narrative Review. Nutrients. 2023 Jan 30;15(3):702. doi: 10.3390/nu15030702. PMID 36771409
- [Background] Bornhorst C, Wijnhoven TM, Kunesova M, Yngve A, Rito AI, Lissner L, Duleva V, Petrauskiene A, Breda J. WHO European Childhood Obesity Surveillance Initiative: associations between sleep duration, screen time and food consumption frequencies. BMC Public Health. 2015 Apr 30;15:442. doi: 10.1186/s12889-015-1793-3. PMID 25924872